CLINICAL TRIAL: NCT00374257
Title: Narrow-Band UVB Phototherapy for Treatment of Oral Chronic Graft-versus-Host Disease
Brief Title: UVB Phototherapy Treatment of Oral Chronic GVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low/slow accrual
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nathaniel Simon Treister, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-054
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2010-03

CONDITIONS: Oral Chronic Graft-versus-host Disease
Keywords: NB-UVB; cGVHD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active intraoral NBUVB therapy (Experimental)
  Interventions: Procedure: Narrow-Band UVB Phototherapy

INTERVENTIONS:
Procedure: Narrow-Band UVB Phototherapy — Performed either two or three times per week for a total of 24 treatments

SUMMARY:
The purpose of this trial is to find out how effective Narrow Band-Ultraviolet Light B (NB-UVB) phototherapy is in treating oral cGVHD. NB-UVB Phototherapy involves exposing the inside of the mouth to light of a particular spectrum (a specific wavelength of light, 311nm) of the ultraviolet band, called NB-UVB. It is known that narrow band ultraviolet light therapy can improve symptoms in patients with skin chronic GVHD.

DETAILED DESCRIPTION:
* At the first visit the following information will be collected about the participant: original diagnosis, the date and type of transplant, transplant conditioning regimen, cGVHD prophylaxis regimen, the time when oral cGVHD was first noticed, specific treatments for oral cGVHD, and any current medications.
* At each visit, and before the participant begins phototherapy treatment, they will answer a series of questions asking about how their mouth feels and what they are able to eat. A clinical examination of the mouth will be performed and recorded and photographs will be taken of the inside of the mouth.
* Participants will then receive phototherapy treatment. This will take approximately three minutes and will involve opening the mouth and closing the eyes. Following phototherapy, the participant will be asked several questions on how they tolerated the treatment. Phototherapy treatments will be done two or three times per week for a total of 24 treatments. After each treatment, if the participant has not experienced any discomfort, the phototherapy dose will be increased following a specific protocol.
* After 24 treatments the participant will have the option to continue phototherapy treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral chronic graft-versus-host disease
* 4 years of age or older
* Stable cGVHD medication regimen for the four weeks prior to study enrollment

Exclusion Criteria:

* New immunomodulatory medications or increasing dosage of current immunomodulatory medications during the four weeks prior to study enrollment
* Concurrent extracorporeal photopheresis.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To clinically evaluate the treatment efficacy of NB-UVB phototherapy in the management of oral cGVHD. | 4 years

SECONDARY OUTCOMES:
To evaluate the convenience, ease of use, tolerability and practicality of NB-UVB phototherapy in this patient population | 4 years
to determine the effective maintenance doses/regimens in participants with good response for long-term management. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel S. Treister, DMD, DMSc, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts